CLINICAL TRIAL: NCT05723393
Title: Sympatholytic Effect of High Thoracic Erector Spinae Plane Block
Brief Title: Sympatholytic Effect of Thoracic ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01-025-01
Record Dates: First submitted 2023-02-02; First posted 2023-02-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 ml T2 ESPB group (Experimental): T2 ESPB group where ESPB is performed at T2 with local anesthetics 20ml
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — fascial plane injection guided by ultrasound

SUMMARY:
The primary endpoint of this study was to identify if erector spinae plane bloock (ESPB) demonstrates any sympatholytic effect.

The secondary endpoint of this study was to compare the changes of PI value between responders and non-responders.

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter. Although the special probe for PI measurement is relatively more expensive compared with ordinary pulse oximetery probes, its benefit as a marker of peripheral perfusion and as an idex for sympathetic stimulation have increased its use progressively.

ESPB can achieve analgesic effect by blocking the ventral and doramal ramus and possibly by diffusion into paravertebral space. In constrast to lumar region, thoracic paravertebral space is very close to the sympathetic chain. Therefore, sympatholytic effect might be achieved by thoracic ESPB. No previous study has demonstrated the sympatholytic effect of ESPB.

ELIGIBILITY:
Inclusion Criteria:

* Complex regional pain syndrome
* Post-thoracotomy pain syndrome
* Cervical foraminal stenosis
* Cervical disc herniation
* Herpes zoster

Exclusion Criteria:

* Pregnacy
* Coagulation abormality
* Previous spine surgery
* Allergy to local anesthetics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Perfusion index changes among 4 times period | baseline, 10minutes after ESPB, 20 minutes after ESPB, 30 minutes after ESPB
  Perfusion index changes after T2 ESPB among 4 times period
Numerical rating scale changes among 3 times period | baseline, 30 minutes after ESPB, 2 weeks after ESPB
  Numerical rating scale changes among 3 times period
Perfusion index ratio at 10 minutes | baseline, 10minutes after ESPB
  Perfusion index ratio at 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ji H Hong, Principal Investigator — Keimyung University
Locations (1):
- Ji Hoon Park, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No